CLINICAL TRIAL: NCT02345200
Title: Body Composition, Muscle Strength and Hormonal Status in Patients With Ataxia Telangiectasia Compared to Healthy Controls
Brief Title: Body Composition and Hormonal Status in Ataxia Telangiectasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Zielen, Prof. Dr. med., Johann Wolfgang Goethe University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BIA_AT2014
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Ataxia Telangiectasia
Keywords: dystrophy; body composition; malnutrition
MeSH Terms: conditions — Ataxia Telangiectasia; Malnutrition | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ataxia telangiectasia (Active Comparator): 26 patients with clinically and/or genetically diagnosed Ataxia telangiectasia will be examined with bioelectrical impedance analysis (BIA), muscle force measurement, calipometry and get a blood draw
  Interventions: Procedure: bioelectrical impedance analysis; Procedure: blood draw
- Healthy subjects (Active Comparator): 26 age and sex matched subjects without any chronic disease or hormone displacement will be examined with bioelectrical impedance analysis (BIA), muscle force measurement, calipometry and get a blood draw
  Interventions: Procedure: bioelectrical impedance analysis; Procedure: blood draw

INTERVENTIONS:
Procedure: bioelectrical impedance analysis — electrophysical measurement that allows to determine the exact composition of single body compartments by producing a magnetic field and detecting the potential difference through the body
Procedure: blood draw — blood samples are taken at 8 am in order to pay attention to the circadian rhythmicity to get a detailed hormonal status

SUMMARY:
Ataxia telangiectasia (A-T) is a rare devastating human recessive disorder characterized by progressive cerebellar ataxia, immunodeficiency, chromosomal instability, and cancer susceptibility. In addition to that, a high percentage of patients show dystrophy, growth retardation and poor weight gain. Nevertheless, there are only a few studies assessing this problem. Aim of the present proposal is to investigate the exact body composition, manual muscle strength and hormonal status in patients with A-T compared to healthy controls matched for gender and age. A pelvic sonography in females was performed in order to evaluate the sexual maturity of their inner genitalia. Tanner score was determined to define the physical development. Every subject received a nutritional diary to review its calorie intake and the quality of diet. The investigators expect that the A-T cohort shows an altered body composition, impaired muscle strength, changed hormonal status concerning the sexual hormones and a delayed physical development compared to healthy controls.

DETAILED DESCRIPTION:
Ataxia telangiectasia (A-T) is a devastating human recessive disorder characterized by progressive cerebellar ataxia, immunodeficiency, chromosomal instability, and cancer susceptibility. In addition to that, a high percentage of patients show dystrophy, growth retardation and poor weight gain. There are only a few studies assessing this problem and the exact variations concerning body composition, muscle strength and hormonal status are widely unknown.

Major factors may be responsible for altered body composition:

1. Immunodeficiency and chronic disease are important influences on growth and physical development. The constantly catabolic situation of A-T patients has a major impact on dystrophy.
2. Due to the progressive cerebellar ataxia most of the patients are bound to wheelchair so that their muscle mass is decreased
3. Impaired muscle strength is related to apraxia, dystonia, contractures and dyskinesia.
4. Low levels of growth hormones (GH). Extracerebellar MRI - lesions in A-T go along with deficiency of the GH axis thus causing nanism.
5. Delayed puberty and physical development suggest an abnormal metabolism in muscle cells
6. There are autopsy reports informing about reduced mass of the adrenal cortex that may be reflected in a lower hormone release of steroid hormones.

The aim of the proposal is to explore the exact body composition, the manual muscle strength, the hormonal status in patients with A-T compared to healthy subjects matched for sex and age. One study visit is performed in all A-T patients and healthy subjects:

* To evaluate weight and length of all subjects
* To analyze the exact structure of single body compartments such as the lean mass, the water compartment or the fat compartment using bioelectrical impedance analysis
* To determine the subcutaneous fat fold thickness using calipometry
* To investigate the nourishment habits and diet detected by nutritional diary
* To analyze the manual muscle strength with a hand dynamometer
* To determine the physical development in the A-T cohort by Tanner scores
* To evaluate stage of sexual development and puberty in female A-T patients by ultrasonic of the inner genitalia
* To get a detailed hormonal status including thyroid-stimulating hormone (TSH), luteinizing hormone (LH), follicle stimulating hormone (FSH), GH, cortisol, DHEAS, estradiol, testosterone, progesterone, insulin like growth factor-binding protein 3 (IGF-BP3), etc in serum blood

ELIGIBILITY:
Inclusion Criteria:

* aim group: clinically and/or genetically diagnosed A-T
* control group: age and sex matched healthy subjects
* age 2-45 years
* written informed consent

Exclusion Criteria:

* age < 2 or > 45 years
* other diseases with influence on the immunosystem (i.e. diabetes mellitus, malignoma, dialysis-dependent renal failure)
* current medication with hormones

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Body mass index | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof. Dr., Principal Investigator — University Childrens´ Hospital Frankfurt

REFERENCES:
- [Background] DUNN HG, MEUWISSEN H, LIVINGSTONE CS, PUMP KK. ATAXIA-TELANGIECTASIA. Can Med Assoc J. 1964 Nov 21;91(21):1106-18. PMID 14229760
- [Background] Schubert R, Reichenbach J, Zielen S. Growth factor deficiency in patients with ataxia telangiectasia. Clin Exp Immunol. 2005 Jun;140(3):517-9. doi: 10.1111/j.1365-2249.2005.02782.x. PMID 15932513
- [Background] Voss S, Pietzner J, Hoche F, Taylor AM, Last JI, Schubert R, Zielen S. Growth retardation and growth hormone deficiency in patients with Ataxia telangiectasia. Growth Factors. 2014 Jun;32(3-4):123-9. doi: 10.3109/08977194.2014.939805. PMID 25060036
- [Background] Kieslich M, Hoche F, Reichenbach J, Weidauer S, Porto L, Vlaho S, Schubert R, Zielen S. Extracerebellar MRI-lesions in ataxia telangiectasia go along with deficiency of the GH/IGF-1 axis, markedly reduced body weight, high ataxia scores and advanced age. Cerebellum. 2010 Jun;9(2):190-7. doi: 10.1007/s12311-009-0138-0. PMID 19898915
- [Background] Cosentino C, Grieco D, Costanzo V. ATM activates the pentose phosphate pathway promoting anti-oxidant defence and DNA repair. EMBO J. 2011 Feb 2;30(3):546-55. doi: 10.1038/emboj.2010.330. Epub 2010 Dec 14. PMID 21157431
- [Background] Baldin AD, Fabbri T, Siviero-Miachon AA, Spinola-Castro AM, de Lemos-Marini SH, Baptista MT, D'Souza-Li LF, Maciel-Guerra AT, Guerra-Junior G. Growth hormone effect on body composition in Turner syndrome. Endocrine. 2011 Dec;40(3):486-91. doi: 10.1007/s12020-011-9504-z. Epub 2011 Jul 1. PMID 21720878
- [Background] Menotta M, Biagiotti S, Bianchi M, Chessa L, Magnani M. Dexamethasone partially rescues ataxia telangiectasia-mutated (ATM) deficiency in ataxia telangiectasia by promoting a shortened protein variant retaining kinase activity. J Biol Chem. 2012 Nov 30;287(49):41352-63. doi: 10.1074/jbc.M112.344473. Epub 2012 Oct 10. PMID 23055520
- [Derived] Pommerening H, van Dullemen S, Kieslich M, Schubert R, Zielen S, Voss S. Body composition, muscle strength and hormonal status in patients with ataxia telangiectasia: a cohort study. Orphanet J Rare Dis. 2015 Dec 9;10:155. doi: 10.1186/s13023-015-0373-z. PMID 26645295